CLINICAL TRIAL: NCT03400072
Title: Adapted Physical Activity in Patients With Resected Pancreatic Cancer (APACaPOp PRODIGE-56 Study): a National Multicenter Randomized Controlled Phase II Trial
Acronym: APACaPOp
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P/2017/317
Record Dates: First submitted 2018-01-09; First posted 2018-01-17 (Actual); Last update posted 2018-11-19 (Actual); Status verified 2018-11

CONDITIONS: Pancreas Cancer; Quality of Life
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Unsupervised APA program (Experimental): usual care plus a 6-month unsupervised APA program
  Interventions: Other: Unsupervised APA program
- Supervised APA program (Experimental): usual care plus a 6-month supervised APA program
  Interventions: Other: Supervised APA program
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Other: Unsupervised APA program — Exercise training program will consist of one supervised demonstration session with the APA professional, thereafter the training will be continued as unsupervised, home-based exercise training sessions.
  Arms: Unsupervised APA program
Other: Supervised APA program — Exercise training program will consist of one supervised demonstration session with the APA professional, thereafter the training will be continued as unsupervised, home-based exercise training sessions; in addition, patients will attend weekly supervised, hospital-based exercise sessions in groups of patients.
  Arms: Supervised APA program

SUMMARY:
Exercise during chemotherapy (CT) is a promising strategy to reduce fatigue and improve health-related quality of life (HRQoL). Exercise may also have beneficial effects on tumor outcome by decreasing insulin resistance, inflammation, and by modulating various pro-tumoral signalling pathways. It has been shown to reduce mortality in breast and colorectal cancer adjuvant setting.

This study aims to explore the effects of adapted physical activity (APA) in patients with resected pancreatic ductal adenocarcinoma (PDAC).

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven PDAC
* Complete macroscopic resection (R0 or R1 resection)
* Patients randomized within 12 weeks of surgery
* No evidence of malignant ascites, liver metastasis, spread to other distant abdominal organs, peritoneal metastasis, spread to extra-abdominal organs
* Sufficient recovery from the operation and fit to take part in the trial
* Able to attend for administration of the adjuvant CT
* ECOG PS 0-2
* Age ≥ 18 years
* Life expectancy > 3 months
* Dated and signed informed consent
* Registration in a national health care system (CMU included).

Exclusion Criteria:

* Macroscopically remaining tumor (R2 resection or TNM stage IV disease)
* Histology other than PDAC
* Cardiovascular, respiratory, psychiatric, musculoskeletal, or neurological condition contra-indicating exercise practice
* Pregnancy or breastfeeding
* Protected adults (individuals under guardianship by court order). Note: participation to another concomitant clinical trial is allowed but the patient must inform and get an authorization from the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Estimated)
Dates: Start 2018-08-03 (Actual); Primary Completion 2022-02 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
M6 Health-Related quality of life (HRQoL) | month 6
  HRQoL will be assessed by the European Organization for Research and Treatment of Cancer quality of life questionnaire (QLQ) C30 at M6, with the following targeted dimensions: global QoL, fatigue, physical functioning, and pain.

CONTACTS AND LOCATIONS:
Overall Officials: Cindy Neuzillet, MD PhD, Principal Investigator — Henri Mondor University Hospital; Pascal Hammel, MD PhD, Principal Investigator — Hôpital Beaujon
Locations (15):
- France (15):
  - CHU de Besançon, Besançon
  - CHU de Brest, Brest
  - Hôpital Beaujon, Clichy
  - Hôpital Henri Mondor, Créteil
  - Hôpital Edouard Herriot, Lyon
  - Hôpital privé Jean Mermoz, Lyon
  - CHR d'Orléans, Orléans
  - Hôpital Cochin, Paris
  - Institut Mutualiste Montsouris, Paris
  - Hôpital Haut-Lévêque, Pessac
  - CHU de Reims, Reims
  - CHU de Rouen, Rouen
  - Institut Curie, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - CHU de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No